CLINICAL TRIAL: NCT07212777
Title: Precisión de la osteotomía Tibial Proximal Con Instrumental Paciente-específico vs técnica Convencional
Brief Title: Precision of Pacient-specific Instrumented Open Wedge High Tibial Osteotomy vs Conventional Technicque
Acronym: AMBE_OR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaga (Other)
Collaborators: Hospital Universitario Virgen de la Victoria (Other)
Responsible Party: Principal Investigator, Dr. Antonio I Cuesta-Vargas, Full Professor, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025999010604889
Record Dates: First submitted 2025-09-23; First posted 2025-10-08 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-09

CONDITIONS: Arthritis (Knee); Varus Knee
Keywords: patient-specific instrumentation; knee osteotomy; Prospective; Randomised Controlled Trial
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional surgery (Active Comparator): Osteotomy using conventional technique
  Interventions: Procedure: Medial Open Wedge Hight Tibial Osteotomy using conventional surgery techniques
- Patient-specific instrumentation (Experimental): Osteotomy using 3D-printed patient-specific instrumentation
  Interventions: Procedure: Medial Open Wedge Hight Tibial Osteotomy using patient-specific instrumentation

INTERVENTIONS:
Procedure: Medial Open Wedge Hight Tibial Osteotomy using patient-specific instrumentation — Medial Open Wedge Hight Tibial Osteotomy using 3D printed patient-specific instrumentation as a guide for the osteotomy
  Arms: Patient-specific instrumentation
Procedure: Medial Open Wedge Hight Tibial Osteotomy using conventional surgery techniques — Conventional Medial Open Wedge Hight Tibial Osteotomy
  Arms: Conventional surgery

SUMMARY:
This study is a randomized clinical trial that will compare two surgical techniques for patients with knee osteoarthritis and varus deformity who are candidates for medial opening wedge high tibial osteotomy. The goal is to evaluate whether using patient-specific 3D-printed surgical guides improves the accuracy of the bone cut compared with the conventional technique performed with anatomical landmarks and fluoroscopy.

A total of 50 adult patients will be randomly assigned to one of two groups: conventional osteotomy or osteotomy assisted by patient-specific instrumentation (PSI). The main outcome is the accuracy of the osteotomy cut, measured by comparing preoperative planning with the postoperative CT scan. Secondary outcomes include leg alignment, surgical time, radiation exposure, complications, and functional recovery assessed with validated questionnaires (KOOS, WOMAC, IKDC, EQ-5D) and gait analysis using depth cameras.

Patients will be followed for up to 12 months after surgery to evaluate clinical and radiological outcomes.

DETAILED DESCRIPTION:
Medial opening wedge high tibial osteotomy is a well-established surgical procedure to correct knee alignment in patients with medial knee osteoarthritis and varus deformity. The accuracy of the bone cut is critical for surgical success. However, conventional techniques performed with anatomical landmarks and fluoroscopy may result in variability and suboptimal correction.

Recent advances in 3D imaging and printing allow the creation of patient-specific surgical guides designed from preoperative CT scans. These guides may improve the accuracy and reproducibility of the osteotomy.

This single-center randomized clinical trial will include 50 adult patients, randomly assigned to undergo conventional osteotomy or osteotomy assisted by patient-specific instrumentation. The main outcome is the accuracy of the osteotomy cut compared with preoperative planning. Secondary outcomes include leg alignment, surgical efficiency, radiation exposure, complications, and functional recovery. Patients will be followed for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent: able to sign informed consent
* Clinical: predominantly medial pain/limitation refractory ≥3-6 months
* Mobility: flexion ≥90º and flexion contracture ≤10º Stability: varus/valgus and pivot-shift ≤ grade 1.
* Radiology:

  * Medial gonarthrosis Ahlbäck I-III with preserved lateral compartment.
  * Patellofemoral Iwano 0-2 without disabling patellofemoral pain.
  * Varus alignment: HKA 4-10°.
  * Predominantly tibial deformity (decreased MPTA; LDFA close to normal) according to planning.
* Anatomy/technical feasibility: proximal tibial morphology suitable for medial opening osteotomy and PSI guide placement.

Exclusion criteria:

* Comorbidity/clinical situations:

  * Inflammatory arthritis (e.g., RA, spondyloarthropathies), unresolved previous joint infection or osteomyelitis.
  * Severe peripheral vasculopathy (ABI <0.7), advanced peripheral neuropathy or Charcot foot.
  * Poorly controlled diabetes (HbA1c >8.5%), advanced renal/hepatic failure (eGFR <30 ml/min/1.73 m²; Child-Pugh B/C).
  * Smoking >20 cigarettes/day without commitment to cessation; active IV drug use or uncontrolled alcoholism.
  * BMI >35 kg/m².
  * Disorder affecting gait (e.g., neurological disease).
  * Inability to walk at a speed of at least 0.8m/s
* Anatomy/radiology

  * Multiplanar deformities not correctable with isolated medial opening tibial valgus osteotomy (e.g., dominant femoral deformity).
  * Severe medial subchondral bone defect or extensive necrosis.
  * Sequelae of proximal tibia fracture or previous ipsilateral HTO that prevent correction or guide use.
* Treatments/medication and logistics

  * Anticoagulation/antiplatelet therapy that cannot be suspended or bridged.
  * Systemic corticosteroids >10 mg/day or high-risk immunosuppressants without possibility of adjustment.
  * Intra-articular infiltration (HA/CS/PRP) within the previous 60 days (respect defined wash-out).
  * Pregnancy.
  * Participation in another interfering trial.
  * Inability to undergo CT (e.g., uncontrollable claustrophobia).
  * Inability to complete ≥12 months of follow-up.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Angular precision in AP and lateral planes | Immediate postoperative period
  Difference between planned and executed angles in AP and lateral planes
Distance to joint line | Immediate postoperative period
  Difference between planned and executed distance between osteotomy cut and and joint line

SECONDARY OUTCOMES:
Postoperative alignment (HKA angle) | Immediate postoperative period
  Difference between planned and achieved hip-knee-ankle angle
Posterior tibial slope (PTS) | Immediate postoperative period
  Difference between planned and achieved tibial slope
Surgical time | Day of surgery
  Duration from skin incision to closure
Number of fluoroscopic images | Day of surgery
  Total intraoperative fluoroscopy shots
Radiation dose | Day of surgery
  Cumulative radiation exposure during surgery (mGy)
Intraoperative complications | Day of surgery
  Events such as hinge fracture or neurovascular injury
Postoperative complications | From surgery to end of 12 month follow-up
  Infection, delayed bone healing, thrombotic events
Reoperation | From surgery to end of 12 month follow-up
  Need for additional surgical intervention
Functional recovery | From surgery to end of 12 month follow-up
  Time to full weight-bearing without assistance
Radiographic consolidation | From surgery until the end of the 12 month follow-up
  Time to radiographic evidence of bone healing
30 Sit to Stand Test | From surgery until the end of the 12 month follow-up
  Amount of sit-to-stands that can be achieved by the patient in a 30 second window
Visual Analog Scale (VAS for pain) | From surgery until the end of the 12 month follow-up
  Range 0-10, where 0 = no pain and 10 = worst imaginable pain. Higher scores indicate worse outcome.
Percentage of patients with a +-2º correction within the planned osteotomy | Immediate postoperative period
  Precision of the alignment of the knee with respect tot he planned osteotomy
Timed-Up-and-Go | From surgery until the end of the 12 month follow-up
  Time that it takes the patient to stand up from a chair and walk 10 meters, turn 180º and return to the starting position
Balance Test (from the Short Physical Performance Battery, SPPB) | From surgery to end of 12 month follow-up
  The balance component of the Short Physical Performance Battery (SPPB) assesses the ability to maintain three standing positions: feet together, semi-tandem, and tandem stand, each for up to 10 seconds. The test is scored from 0 to 4, where 0 = unable to hold any position, and 4 = able to hold the tandem position for 10 seconds. Higher scores indicate better balance performance.
Knee injury and Osteoarthritis Outcome Score (KOOS) | From surgery to end of 12 month follow-up
  Each subscale scored from 0-100, where 0 = extreme problems and 100 = no problems. Higher scores indicate better outcome.
International Knee Documentation Committee (IKDC) Subjective Knee Evaluation Form | From surgery to end of 12 month follow-up
  Score range 0-100, where 0 = worst knee function and 100 = no limitations. Higher scores indicate better outcome.
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | From surgery to end of 12 month follow-up
  Scored 0-96, where higher scores indicate worse pain, stiffness, and physical function.
EuroQol 5 Dimensions Questionnaire (EQ-5D-5L) | From surgery to end of 12 month follow-up
  Index score range usually from -0.59 (worst health state) to 1 (perfect health); higher scores indicate better quality of life.
Lower Limb Functional Index (LLFI) | From surgery to end of 12 month follow-up
  Patient-reported questionnaire that measures lower limb functional status. It consists of 25 items scored as "yes" (1 point), "sometimes" (0.5 points), or "no" (0 points). The raw score is summed and converted to a percentage (0-100). Higher scores indicate greater disability, while lower scores indicate better functional status. Ranges from 0-100. Higher scores mean a worse outcome.
Foot Health Status Questionnaire (FHSQ) | From surgery to end of 12 month follow-up
  Patient-reported questionnaire assessing foot health across several domains: pain, function, footwear, and general foot health. Each domain score is transformed to a 0-100 scale. Higher scores indicate better foot health and function. Range: 0-100 for each domain. Higher scores mean a better outcome.
Foot Function Index (FFI) | From surgery to end of 12 month follow-up
  Patient-reported measure assessing foot pain, disability, and activity limitation. Contains 23 items scored on a visual analog scale (0-10). The total score is normalized to a 0-100 scale. Higher scores indicate greater pain, disability, and activity limitation. Range: 0-100. Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio I Cuesta-Vargas, Prof., PhD, Principal Investigator — Universidad de Málaga; Juan Miguel Gómez-Palomo, PhD, Principal Investigator — Hospital Universitario Virgen de la Victoria
Locations (1):
- Hospital Universitario Virgen de la Victoria de Málaga, Málaga, Málaga, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Studenski S, Perera S, Patel K, Rosano C, Faulkner K, Inzitari M, Brach J, Chandler J, Cawthon P, Connor EB, Nevitt M, Visser M, Kritchevsky S, Badinelli S, Harris T, Newman AB, Cauley J, Ferrucci L, Guralnik J. Gait speed and survival in older adults. JAMA. 2011 Jan 5;305(1):50-8. doi: 10.1001/jama.2010.1923. PMID 21205966
- [Result] Jacquet C, Sharma A, Fabre M, Ehlinger M, Argenson JN, Parratte S, Ollivier M. Patient-specific high-tibial osteotomy's 'cutting-guides' decrease operating time and the number of fluoroscopic images taken after a Brief Learning Curve. Knee Surg Sports Traumatol Arthrosc. 2020 Sep;28(9):2854-2862. doi: 10.1007/s00167-019-05637-6. Epub 2019 Jul 27. PMID 31352498
- [Result] Pang R, Jiang Z, Xu C, Shi W, Zhang X, Wan X, Bahat D, Li H, Senatov F, Bulygina I, Wang H, Zhang H, Li Z. Is Patient-Specific Instrumentation Accurate and Necessary for Open-Wedge High Tibial Osteotomy? A Meta-Analysis. Orthop Surg. 2023 Feb;15(2):413-422. doi: 10.1111/os.13483. Epub 2022 Dec 30. PMID 36585795
- [Result] Zhu X, Qian Y, Liu A, Xu P, Guo JJ. Comparative outcomes of patient-specific instrumentation, the conventional method and navigation assistance in open-wedge high tibial osteotomy: A prospective comparative study with a two-year follow up. Knee. 2022 Dec;39:18-28. doi: 10.1016/j.knee.2022.08.013. Epub 2022 Sep 14. PMID 36115179
- [Result] Cerciello S, Ollivier M, Corona K, Kaocoglu B, Seil R. CAS and PSI increase coronal alignment accuracy and reduce outliers when compared to traditional technique of medial open wedge high tibial osteotomy: a meta-analysis. Knee Surg Sports Traumatol Arthrosc. 2022 Feb;30(2):555-566. doi: 10.1007/s00167-020-06253-5. Epub 2020 Sep 10. PMID 32910222
- [Result] Carey EG, Kamath AF, Vidal AF, Frush T, Alaia M, Baldwin RB, Ranawat A. Assessing the Impact of Patient-Specific Instrumentation and Fixation on Accuracy and Radiation Exposure in a Cadaveric Model of Medial Opening-Wedge High Tibial Osteotomy. Orthop J Sports Med. 2025 Jan 28;13(1):23259671241285430. doi: 10.1177/23259671241285430. eCollection 2025 Jan. PMID 39881858
- [Result] Miao Z, Li S, Luo D, Lu Q, Liu P. The validity and accuracy of 3D-printed patient-specific instruments for high tibial osteotomy: a cadaveric study. J Orthop Surg Res. 2022 Jan 29;17(1):62. doi: 10.1186/s13018-022-02956-2. PMID 35093132
- [Result] Chaouche S, Jacquet C, Fabre-Aubrespy M, Sharma A, Argenson JN, Parratte S, Ollivier M. Patient-specific cutting guides for open-wedge high tibial osteotomy: safety and accuracy analysis of a hundred patients continuous cohort. Int Orthop. 2019 Dec;43(12):2757-2765. doi: 10.1007/s00264-019-04372-4. Epub 2019 Jul 5. PMID 31273430
- [Result] Donnez M, Ollivier M, Munier M, Berton P, Podgorski JP, Chabrand P, Parratte S. Are three-dimensional patient-specific cutting guides for open wedge high tibial osteotomy accurate? An in vitro study. J Orthop Surg Res. 2018 Jul 9;13(1):171. doi: 10.1186/s13018-018-0872-4. PMID 29986731
- [Result] Jones GG, Jaere M, Clarke S, Cobb J. 3D printing and high tibial osteotomy. EFORT Open Rev. 2018 May 21;3(5):254-259. doi: 10.1302/2058-5241.3.170075. eCollection 2018 May. PMID 29951264
- [Result] Stimolo D, Leggieri F, Matassi F, Barra A, Civinini R, Innocenti M. Learning curves for high tibial osteotomy using patient-specific instrumentation: a case control study. Innov Surg Sci. 2024 Jul 3;9(3):123-131. doi: 10.1515/iss-2024-0007. eCollection 2024 Sep. PMID 39309194